CLINICAL TRIAL: NCT01719809
Title: A Prospective Evaluation of the Effect of Training on Eye Drop Administration in Glaucoma Subjects Who Have Difficulties Properly Instilling Eye Drops
Brief Title: An Evaluation of the Ability to Train Established Glaucoma Patients Who Have Difficulty in Drop Instillation
Status: Terminated | Type: Observational
Why Stopped: Enrollment Goals not met
Sponsor: Robin, Alan L., M.D. (Individual)
Responsible Party: Principal Investigator, Adam C. LePosa, Adam C. LePosa, O.D, Robin, Alan L., M.D.
Other Study IDs: ALR 0054
Record Dates: First submitted 2012-10-25; First posted 2012-11-01 (Estimated); Last update posted 2017-04-12 (Actual); Status verified 2017-04

CONDITIONS: Glaucoma; Ocular Hypertension
Keywords: Glaucoma; Eye Drop; Eye Drop Technique; Training; Instilling Eye Drops
MeSH Terms: conditions — Glaucoma; Ocular Hypertension

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This is a prospective, observational, single-center study. Patients with at least 3 months of experience using topical medications for glaucoma and who state that they administer their own eye drops will be recruited. Subjects will be videotaped instilling a sterile artificial eye drop, will be identified at the time of a regularly scheduled exam. If the patient can get a drop onto the eye and also not touch their lids or ocular surface with the eye drop bottle, the subject will be thanked but not enrolled. All other patients who agree to participate will be enrolled. Upon completion of videotaped instillation of an eye drop, each enrolled patient will be shown a video demonstrating an instillation technique and will be given an instructional handout highlighting a proper drop instillation technique. If necessary, an instillation technique will be demonstrated to them by an investigator or trained personnel.

A patient will be identified as properly instilling a drop if they satisfy the following criteia:

They are able to instill one (and only one) drop to the ocular surface or lower fornix without allowing the bottle touch the adnexa, eyelid, eye lashes or eye.

All patients routinely return between 3 and 6 months. At this regularly scheduled visit,the investigator or trained personnel would direct the patient to instill an eye drop into the study eye.Additionally, the short glaucoma self-efficacy questionnaire will be re-administered.

All of the video-recordings of participants' eye drop instillation techniques will be reviewed and assessed using a standard checklist. Their ability to administer an eye drop after training will be compared to baseline.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or older
* Patients currently using topical ocular antihypertensive medications at the time of enrollment in at least one eye, and who have been using these drops consistently for a period of at least three months prior to enrollment.
* Patients with primary open angle glaucoma, pigmentary glaucoma, exfoliation glaucoma, ocular hypertension, normal-tension glaucoma, neovascular glaucoma, uveitic glaucoma and chronic narrow angle glaucoma.
* Patients CAN be enrolled even if they have co-existing morbidities such as Parkinson's Disease or arthritis

Exclusion Criteria:

* Patients who do not instill their own eye drops
* Patients who are not expected to still be using topical antihypertensive medications at the time of study follow-up
* Patients with no light perception vision
* Patients with a history of adverse reaction to artificial tears or any component of artificial tears
* Patients who have a typical follow-up period of greater than 6 months
* Patients who have not completed a Humphrey Visual Field C24-2 or C10-2 within 7 months of enrollment or study exit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Private Ophthalmology Office (Specialty-Glaucoma)
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2012-10; Primary Completion 2015-06 (Actual); Study Completion 2015-06-01 (Actual)

PRIMARY OUTCOMES:
Ability to administer an eye drop according to our criteria, as outlined in our study summary. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Adam C LePosa, OD, Principal Investigator — Alan L. Robin, MD, PA
Locations (1):
- Alan L. Robin, MD, PA, Baltimore, Maryland, United States